CLINICAL TRIAL: NCT07195955
Title: The Effect of Cold Spray Application in Reducing Pain and Ecchymosis in Patients Receiving Low Molecular Weight Heparin Prophylaxis After Orthopedic Surgery
Brief Title: Cold Spray for Pain and Ecchymosis After Anticoagulant Prophylaxis in Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Şükriye ŞAHİN, Research Assistant, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024/07.40.
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Nursing Care; Cold Application; Pain; Ecchymosis
Keywords: nursing care; cold application; pain; ecchymosis
MeSH Terms: conditions — Pain; Ecchymosis

STUDY DESIGN:
Intervention Model Description: The study was conducted experimentally with a pre-test and post-test control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study employed a single-blind design. To prevent bias in the analysis of the research data, blinding was also applied to the outcomes assessor and statistician. The care provider and researcher in the study were composed of different individuals. When coding the research data, the study groups were coded as A and B, preventing the statistician from knowing which letter represented which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Spray Application (Experimental): In patients who receive standard and routine subcutaneous low molecular weight heparin (LMWH) prophylaxis after orthopedic surgery, cold spray is applied to the injection site before this injection.
  Interventions: Other: Cold Spray Application
- Standart (Routine) Care (No Intervention): This injection is administered without cold application to patients receiving standard and routine subcutaneous low molecular weight heparin (LMWH) prophylaxis after orthopedic surgery.

INTERVENTIONS:
Other: Cold Spray Application — A cold spray is applied to the skin at the planned injection site immediately before LMWH administration to reduce pain and ecchymosis.
  Arms: Cold Spray Application

SUMMARY:
Heparin is a widely used anticoagulant for thrombosis prevention, and low molecular weight heparin (LMWH) has become the preferred option due to its higher bioavailability, strong antithrombotic effect, and lower risk of complications. However, subcutaneous LMWH injections-commonly administered in the abdomen, arm, or thigh-often cause local side effects such as pain, ecchymosis, and hematoma. The incidence of ecchymosis after injection ranges between 26-89%, and various factors such as injection site, needle size, injection duration, and techniques can influence these outcomes. Cold application is frequently used to reduce injection-related pain and bruising by inducing vasoconstriction, decreasing nerve conduction, and increasing pain tolerance.

In orthopedic surgery patients, limited injection sites due to dressings, casts, or splints may increase the risk of repeated bruising and pain. Although cold compresses have been studied in reducing injection-related complications, no research has evaluated the effect of cold spray prior to LMWH administration in this patient group. Therefore, standardized studies are needed to determine whether cold spray is an effective, practical alternative for reducing pain and ecchymosis following LMWH prophylaxis after orthopedic surgery.

DETAILED DESCRIPTION:
Heparin is an anticoagulant used in the surgical prevention of thrombosis and can prevent and treat venous thrombosis by rapidly achieving its anticoagulant effects. Low molecular weight heparin (LMWH), a relatively new anticoagulant developed in the 1970s, has the advantages of high bioavailability, potent antithrombotic effect, a low risk of heparin-induced thrombocytopenia, and fewer bleeding side effects. Therefore, LMWH is increasingly used in clinical practice. Venous thromboembolism is a common complication during and after hospitalization in medical and surgical patients, including orthopedic patients. Without any prophylaxis, the incidence of fatal pulmonary embolism in hospitalized patients is 0.1-0.8% after elective general surgery, 2-3% after elective hip replacement, and 4-7% after hip fracture surgery. Therefore, patients receive heparin for several days or weeks from hospital admission until discharge.

Nurses, in their therapeutic role, administering medications is one of the most fundamental nursing functions requiring knowledge and skill.The basis of medication administration is to ensure patient safety, enhance the beneficial effects of the medication, prevent complications, and increase individual satisfaction and comfort.

The primary route of administration for low molecular weight heparin (LMWH) is subcutaneous injection into the abdominal area, midline of the triceps muscle, or lateral thigh. This method is preferred due to its easy accessibility and slow absorption of the medication. However, local side effects such as pain, ecchymosis (26.6%-88.9%), hematoma (40%-88%), and, in rare cases, tissue sclerosis can occur. Post-injection ecchymosis often occurs between 48 and 72 hours. Factors affecting the pain and bruising caused by subcutaneous injection of LMWH may include injection time; different injection sites; LMWH dose; needle size; slow delivery of heparin to tissues; use of the aspiration airlock technique; and cold application. Cold application has been frequently used to prevent injection-related pain and ecchymosis. In cold applications, when the skin temperature drops to 15 °C, vasoconstriction develops in superficial vessels, and vasodilation develops as the temperature drops even lower. Cold application reduces muscle spasm by slowing down the conduction properties of peripheral nerves and increases pain tolerance. Additionally, vasoconstriction resulting from cold application can reduce blood flow to the tissue, reducing bruising and hematoma formation.

After orthopedic surgery, patients are applied a dressing, bandage, cast, or splint, and post-traumatic bruising or ecchymosis can occur in many areas of the skin. Therefore, injection sites are limited, making rotation between these areas difficult. Using the same area can lead to the formation of new ecchymosis and increased pain sensitivity in the area. There are no studies in the literature on the effects of cold spray applied before SC LMWH application after orthopedic surgery. A more standardized and practical study is needed to evaluate the effects of cold spray on pain and ecchymosis, which can be achieved with cold compresses instead of cold compresses.

ELIGIBILITY:
Inclusion Criteria:

Patients who are:

* 18 years of age or older
* Receiving 1 x 0.4 ml anticoagulant therapy
* Are on the first day of LMWH therapy
* Have no infection, scar tissue, lipodystrophy, or incision at the injection site
* Have not received any other parenteral therapy at the injection site
* Are not allergic to cold or heparin
* Volunteer to participate in the study

Exclusion Criteria:

* Patients were excluded from the study if they were: • Pregnant, • Had any acute or chronic coagulation disorder or hematological disease,

  * Had a subcutaneous injection into the same area 24 hours prior,
  * Wanted to withdraw from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-02-03 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Immediately after each LMWH injection.
  Pain intensity at the injection site will be measured using the Visual Analog Scale (VAS). 10-cm VAS scale (0 = no pain, 10 = worst possible pain).
Ecchymosis Area | 48 and 72 hours after injection.
  The size of ecchymosis at the injection site will be measured using the Opsite-Flexigrid transparent film. Area calculated in cm² by tracing the ecchymosis on the grid.

CONTACTS AND LOCATIONS:
Overall Officials: YASEMİN ÖZHANLI, Assist.Prof, Study Director — Kocaeli University; HATİCE MERVE ALPTEKİN, Research Assistant, Study Chair — Kocaeli University; ALİ OSMAN ALTUNTAŞ, Student, Study Chair — Kocaeli University
Locations (1):
- Kocaeli University, Köseköy, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ekanayake C, Gamage JCPH, Mendis P, Weerasinghe P. Revolution in orthopedic immobilization materials: A comprehensive review. Heliyon. 2023 Feb 16;9(3):e13640. doi: 10.1016/j.heliyon.2023.e13640. eCollection 2023 Mar. PMID 36915506
- [Result] Sendir M, Buyukyilmaz F, Celik Z, Taskopru I. Comparison of 3 methods to prevent pain and bruising after subcutaneous heparin administration. Clin Nurse Spec. 2015 May-Jun;29(3):174-80. doi: 10.1097/NUR.0000000000000129. PMID 25856035
- [Result] Erek Kazan, E. (2021). Hot and cold applications. In M. Kara Kaşıkçı & E. Akın (Eds.), Fundamentals of nursing: Concepts, principles, practices (1st ed., pp. 492-515). Istanbul Medical Bookstores.
- [Result] Lafcı, D. (2021). Hot and cold applications. In N. Sabuncu, S. Erkal İlhan, & Z. Koç (Eds.), Fundamentals of nursing care: Concepts, principles, practices (pp. 801-823). Alter Publishing.
- [Result] Çalışkan, N. (2021). Hot and cold applications. In T. Atabek Aşti & A. Karadağ (Eds.), Fundamentals of nursing: From knowledge to practice - Concepts, principles, skills (2nd ed., pp. 567-586). Akademi Publishing.
- [Result] Altaie, A. H., AbdulRazzaq, H. A., & Abd Al-hadi, A. (2013). Dose effect and risk factors on the severity of enoxaparin bruising side effect. International Journal of Clinical Pharmacy, 35(5), 950.
- [Result] Palese A, Aidone E, Dante A, Pea F. Occurrence and extent of bruising according to duration of administration of subcutaneous low-molecular-weight heparin: a quasi-experimental case-crossover study. J Cardiovasc Nurs. 2013 Sep-Oct;28(5):473-82. doi: 10.1097/JCN.0b013e3182578b87. PMID 22760174
- [Result] Bayram SB, Gulnar E, Caliskan N, Kosucu P, Bektas O, Bayram A, Aksoy F. The Effect of Two Types of Subcutaneous Heparin Injections on Pain, Ecchymosis, Hematoma and Drug Absorption: A Quasi-Experimental Study. J Eval Clin Pract. 2025 Feb;31(1):e14266. doi: 10.1111/jep.14266. PMID 39660578
- [Result] Amaniyan S, Varaei S, Vaismoradi M, Haghani H, Sieloff C. Effect of local cold and hot pack on the bruising of enoxaparin sodium injection site: a randomized controlled trial. Contemp Nurse. 2016 Feb;52(1):30-41. doi: 10.1080/10376178.2016.1190289. Epub 2016 Jun 5. PMID 27207493
- [Result] Karadag S, Aydinli A, Yilmaz C, Tutar N. Effect of cold application and compression on pain and bruising in subcutaneous heparin injection. J Vasc Nurs. 2023 Mar;41(1):22-26. doi: 10.1016/j.jvn.2023.01.002. Epub 2023 Jan 17. PMID 36898801
- [Result] Tosun, H. (2019). Medication management: Oral and local drug administration. In T. Atabek Aşti & A. Karadağ (Eds.), Fundamentals of nursing: From knowledge to practice - Concepts, principles, skills. Akademi Publishing.
- [Result] Taylor, C., Lynn, P., & Bartlett, J. (2018). Fundamentals of nursing: The art and science of person-centered care (pp. 59-380). Wolters Kluwer.
- [Result] Duruk, N. (2023). Nursing functions and roles. In M. Kara Kaşıkçı & E. Akın (Eds.), Fundamentals of nursing: Concepts, principles, practices (pp. 11-17). Istanbul Medical Bookstores.
- [Result] Flevas DA, Megaloikonomos PD, Dimopoulos L, Mitsiokapa E, Koulouvaris P, Mavrogenis AF. Thromboembolism prophylaxis in orthopaedics: an update. EFORT Open Rev. 2018 Apr 27;3(4):136-148. doi: 10.1302/2058-5241.3.170018. eCollection 2018 Apr. PMID 29780621
- [Result] Hallan SS, Kaur V, Jain V, Mishra N. Development and characterization of polymer lipid hybrid nanoparticles for oral delivery of LMWH. Artif Cells Nanomed Biotechnol. 2017 Dec;45(8):1631-1639. doi: 10.1080/21691401.2016.1276920. Epub 2017 Jan 10. PMID 28071140
- [Result] Wang H, Guan J, Zhang X, Wang X, Ji T, Hou D, Wang G, Sun J. Effect of Cold Application on Pain and Bruising in Patients With Subcutaneous Injection of Low-Molecular-Weight Heparin: A Meta-Analysis. Clin Appl Thromb Hemost. 2020 Jan-Dec;26:1076029620905349. doi: 10.1177/1076029620905349. PMID 32372652